CLINICAL TRIAL: NCT05893303
Title: Effect of Proprioceptive Neuromuscular Facilitation (PNF) Techniques on Balance and Gait Characteristics of Elderly People with Scapular Disposition: a Randomized Controlled Trial
Brief Title: Effect of Proprioceptive Neuromuscular Facilitation Techniques on Elderly People with Scapular Disposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK022.04
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-07

CONDITIONS: Geriatric Rehabilitation; Scapular Dyskinesis
Keywords: Geriatric Rehabilitation; Scapular Disposition; Balance; Posture; Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PNF Technique Group (Experimental): Participants in this group will receive PNF techniques and gait training 3 times per week for 8 weeks
  Interventions: Other: 1st Group
- Gait Training Group (Active Comparator): Participants in this group will receive only gait training 3 times per week for 8 weeks
  Interventions: Other: 2nd Group

INTERVENTIONS:
Other: 1st Group — 1st group is going to undergo scapula-oriented PNF techniques (diagonal) which are anterior elevation and posterior depression - posterior elevation and anterior depression with 20 repetitions with rhythmic initiation and repeated contractions facilitation techniques during all patterns. In addition to PNF techniques, gait training is going to be applied as standing with balance exercises (15 repetitions) as well as specific exercises for the stance and swing phases of the gait which are; stepping forward and sideways (15 repetitions), and gait education (walking 3 lapses within 2 meters parallel bar)
  Arms: PNF Technique Group
Other: 2nd Group — 2nd group is going to undergo only gait training and balance exercises (15 repetitions) as well as specific exercises for the stance and swing phases of the gait which are; stepping forward and sideways (15 repetitions), and gait education (walking 3 lapses within 2 meters parallel bar)
  Arms: Gait Training Group

SUMMARY:
Proprioceptive neuromuscular facilitation (PNF) has been defined as a comprehensive rehabilitation approach focusing on a motor learning effect, especially in the elderly. Therefore, PNF can be an effective treatment method for our purpose which is to analyze if PNF techniques improve balance and gait characteristics in elderly with scapular disposition and to determine the difference when used with the gait education

DETAILED DESCRIPTION:
Participants will be randomly divided into 2 groups. Scapular PNF techniques in addition to gait training will be applied to the 1st group for 8 weeks, and only gait training exercises will be applied to the 2nd group for 8 weeks. Individuals will be evaluated in detail at the beginning, and end of the study, and after 3 months as a follow-up evaluation. For the assessment of scapular disposition, the Visual Scapular Disposition Test and Lateral Scapular Slide Test will be applied. Walking Speed will be evaluated with a dedicated area by measuring the distance. The Modified Dynamic Gait Index will be used for measuring the ability of the participant to maintain walking balance while responding to different task demands. For fall risks and functional mobility Timed Up and Go Test and Falls Efficacy Scale will be used. For balance assessment Berg Balance Scale and Functional Reach Test. For assessment of the quality of life, SF-36 will be used. Posture will be assessed with a dedicated application called PostureCo

ELIGIBILITY:
Inclusion Criteria:

* Having scapular disposition (Patients will be determined after the visual scapular disposition test and lateral scapular slide test)
* With no injuries
* Able to walk without any assistive devices
* To be able to read and write in Turkish

Exclusion Criteria:

* Having a musculoskeletal or neurological problem that causes issues with applying the intervention.
* Any orthopedic, neurological, cardiac, vestibular, visual, or psychiatric impairment which would not allow them to perform
* Had physiotherapy during the past 3 months

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Visual Scapular Disposition Test | 5 minutes
  During the visual scapular disposition test, patients will be asked to perform bilateral shoulder elevation movements and scapular movements will be observed in order to determine scapular dyskinesia
Lateral Scapular Slide Test | 5 minutes
  During the lateral scapular slide test, patients will be evaluated in 3 different arm positions while standing. at each position, special measurements of the scapula will be taken with measurement tape. If the difference between measurements in the same position is more than 1.5 centimeters (cm), the patient will be recorded as having scapular dyskinesia
Walking Speed | 5 minutes
  Participants normal walking speed measurement will be taken by asking patient to walk a dedicated 15m line and normal walking speed will be measured after 3 repetitions average time calculated
Modified Dynamic Gait Index (mDGI) | 10 minutes
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions.
Timed Up and Go Test | 5 minutes
  The timed "get up and walk" test is the basic functional mobility test for the elderly which they will be asked to stand up from a regular chair, walk 3 meters, turn and walk back to the chair and sit.
Berg Balance Scale | 5 minutes
  Berg Balance Scale (BDI) is generally used to measure balance performance in elderly patients. It is effective in assessing postural control and predicting fall risk.
Functional Reach Test | 5 minutes
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for assessing dynamic balance in one simple task. It will be done in the standing position, by measuring the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support, and this information is correlated with the risk of falling
Falls Efficacy Scale | 5 minutes
  The Falls Efficacy Scale is a short, easy to administer tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity.
PostureCO | 5 minutes
  PostureCo, Inc. is a technology company focusing on posture and movement analysis, it takes the data for the posture and movements. A special posture application for mobile phones will be used to determine postural sway. Data will be collected by scanning each patient and analyzing the posture.
SF-36 | 5 minutes
  The 36-item Short Form (SF-36) is a commonly used questionnaire for measuring health-related quality of life. Each patient will be asked to answer the questions in order to get the results for the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Belgen Kaygisiz, PT, PhD, Principal Investigator — European University of Lefke
Locations (1):
- Fizyomorfo Fizyoterapi Rehabilitasyon ve Saglikli Yasam Merkezi, Güzelyurt, TRNC, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No